CLINICAL TRIAL: NCT03073512
Title: The Role of Fetal Ductus Arteriosus in Predicting Spontaneous Preterm Birth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to locate the resources necessary to complete participant recruitment.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-038
Record Dates: First submitted 2017-02-15; First posted 2017-03-08 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound examination (Other): Participants will undergo an ultrasound examination at 32 weeks gestation.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Participants will undergo ultrasound examination at 32 weeks gestation

SUMMARY:
Preterm birth still remains a major cause of perinatal morbidity and mortality worldwide. The exact mechanism stimulating term and preterm births in humans is still unknown. Prostaglandins, by mediating cervical ripening and early stimulation of myometrial contractions, are likely to play a major role in the parturition process. Much of the unique fetal circulation is facilitated by the ductus arteriosus. Patency of the ductus arteriosus in utero is primarily maintained via prostaglandins which are highly expressed by smooth muscle cells located in the media of the ductus arteriosus. The primary objective of this study is to prospectively assess whether any changes in the fetal ductus arteriosus parameters exist at 32 weeks' gestation. The secondary objective is to investigate whether there is an association between the ductus arteriosus parameters and the time to delivery interval at 32 weeks' gestation.

DETAILED DESCRIPTION:
The rationale is to assess whether physiological responses that occur around the time of delivery, in both the mother and the fetus (elevated prostaglandins level), can be quantified using ultrasound of the fetal ductus arteriosus.

Whether or not the ductus arteriosus plays an active physiological role in the initiation of parturition is unknown. Since prostaglandins are physiologically highly expressed within the fetal ductus arteriosus and also linked to some critical steps throughout parturition, it is hypothesized that structural and doppler flow pattern variations of the ductus arteriosus exist in the period surrounding the birth. These changes might occur before or after the intrinsic rise of prostaglandins and could be quantified using prenatal ultrasound of the fetal ductus arteriosus.

Identifying new physiological based variables that can assist in predicting the onset of labour, especially surrounding preterm birth, as the one suggested in the current study, is thus of great importance and may provide invaluable information into the overall future care and decision making during pregnancy, especially around the time of delivery. It may assist in creating future recommendations for pregnant women and improved healthcare standards during the delivery process.

ELIGIBILITY:
Inclusion criteria:

* Low risk singleton pregnancy at 32 weeks gestation.

Exclusion criteria:

* Smoking
* Underlying cardiac or respiratory illness
* Fetal growth restriction
* Medicated gestational hypertension or evolving preeclampsia
* Gestational diabetes controlled with insulin or oral medications
* Use of steroids for lung maturation in the current pregnancy
* Known major congenital anomalies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Fetal ductus arteriosus changes | 32 weeks gestation
  To prospectively assess any changes in blood flow in the fetal ductus arteriosus at 32 weeks' gestation.

SECONDARY OUTCOMES:
Time to delivery | 32 weeks gestation to delivery
  To investigate whether there is an association between the ductus arteriosus parameters and the time to delivery interval at 32 weeks' gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No